CLINICAL TRIAL: NCT03099018
Title: Comparison of Two Rapid Antigen Detection Tests for the Detection of Group-A Streptococcal Pharyngitis in Children
Status: Completed | Type: Observational
Sponsor: University Hospital, Geneva (Other)
Collaborators: Quidel Corporation (Industry)
Responsible Party: Principal Investigator, Laurence Lacroix, MD, Pediatric Emergency Physician, University Hospital, Geneva
Other Study IDs: 13-248
Record Dates: First submitted 2017-03-28; First posted 2017-04-04 (Actual); Last update posted 2017-04-17 (Actual); Status verified 2017-04

CONDITIONS: Pharyngitis
Keywords: GAS; pharyngitis; children; RADT
MeSH Terms: conditions — Pharyngitis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: Sofia Strep A FIA — Patients who presented with sore throat will be performed throat swab for the new fluorescent immunoasssay (Sofia Strep A FIA), for a standard RADT (Alere Testpack Strep A) and for culture and backup PCR in case of discrepant results.

SUMMARY:
Group A streptococcal (GAS) pharyngitis in children represents a frequent diagnostic challenge in pediatric emergency departments, since isolated signs and clinical prediction rules are insufficient to accurately discriminate between GAS and non GAS infections. Rapid antigen detection tests (RADTs) therefore remain essential, simple and rapid tools, allowing for rapid GAS identification and prompt antibiotic prescription. However, their sensitivity is not optimal. The aim of the present study is to test the accuracy of a new fluorescent immunoassay (Sofia Strep A FIA) using the optical technology for GAS detection in children 3-15 years old with pharyngitis, compared to a standard RADT, using throat culture as the gold standard (or PCR for discrepant results, i.e. negative culture with any positive RADT).

ELIGIBILITY:
Inclusion Criteria:

* Patient age between 3 and 15 years
* Clinical diagnosis of pharyngitis
* McIsaac score ≥2

Exclusion Criteria:

* Antibiotic treatment in the two weeks preceding the consultation

Ages: 3 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children 3 to 15 years old presenting to the PED with pharyngitis and Mc Isaac score ≥ 2
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2014-06 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy of the new Sofia Strep A FIA test in children with pharyngitis | 1 hour
  Comparison of the sensitivity and specificity of two rapid tests (Sofia StrepA FIA and Alere Testpack Strep A) using standard throat culture as reference.

SECONDARY OUTCOMES:
Diagnostic accuracy of the new Sofia Strep A FIA test in children with pharyngitis stratified on the pretest probability of GAS infection (according to McIsaac scores) | 1 hour
  sensitivity and specificity of the two tests in relationship to the pretest-probability of GAS infection as measured by the McIsaac score

CONTACTS AND LOCATIONS:
Overall Officials: Laurence Lacroix, MD, Principal Investigator — University Hospital, Geneva

IPD SHARING:
Plan to Share IPD: No